CLINICAL TRIAL: NCT07278219
Title: The Effect of Balint Approach Group Intervention on Burnout and Communication Skills in Nurses
Brief Title: Balint Approach Group Intervention
Acronym: Balint Group
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuksek Ihtisas University (Other)
Responsible Party: Principal Investigator, Reyhan Dogan, Assistant Professor of Psychiatric Nursing, Yuksek Ihtisas University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: E-10333602-050.04-280361
Record Dates: First submitted 2025-11-28; First posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Burnout; Communication Skills; Psychosocial Well-being
Keywords: burnout; Communication skills; nursing
MeSH Terms: conditions — Burnout, Psychological

STUDY DESIGN:
Intervention Model Description: This study used a two-arm parallel assignment model in which participants were randomly allocated to either the intervention group or the control group in a 1:1 ratio. Both groups were followed concurrently, and outcome assessments were conducted at identical time points (baseline, post-intervention, 1-month follow-up, and 3-month follow-up). No crossover between groups occurred
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm Title: Balint-Based Group Intervention (Experimental): Participants in this arm received a Balint-based group intervention consisting of six weekly online sessions, each lasting 45-50 minutes. Sessions followed the structure recommended by the International Balint Federation, including case presentation, exploration, group discussion, feedback, and closing phases. The intervention was delivered by two psychiatric nursing academics trained in psychotherapy techniques. The group was conducted as a closed group, and sessions were scheduled according to nurses' shift patterns
  Interventions: Behavioral: Balint Approach Group Intervention
- Arm Title → Control Group (No Intervention) (No Intervention): Participants in this arm continued their routine work schedules and did not receive any additional training, counseling, or psychosocial intervention during the study period. Data collection was performed at the same time points as the intervention group (baseline, post-intervention, 1-month follow-up, and 3-month follow-up). After the study was completed, the control group was informed about the intervention

INTERVENTIONS:
Behavioral: Balint Approach Group Intervention — A Balint-based group intervention consisting of six weekly online sessions lasting 45-50 minutes. Sessions followed the structure recommended by the International Balint Federation, including case presentation, exploration, group discussion, feedback, and closing phases. The intervention was delivered by two psychiatric nursing academics trained in psychotherapy techniques. The group was conducted as a closed group, and sessions were scheduled according to participants' shift patterns
  Other Names: Balint-Based Group Intervention
  Arms: Arm Title: Balint-Based Group Intervention

SUMMARY:
This randomized controlled trial evaluated the effect of a Balint-based group intervention on burnout and communication skills among nurses. Burnout is a common outcome of prolonged exposure to workplace stressors and can weaken nurses' empathy, emotional regulation, and therapeutic communication abilities. Balint groups are reflective, structured sessions that focus on understanding the emotional and relational aspects of challenging patient-nurse interactions. These groups provide a safe environment for nurses to explore their thoughts and feelings, enhance self-awareness, and improve interpersonal effectiveness.

The study used a two-arm parallel-group randomized controlled design with pre-test and post-test measurements and follow-up assessments at one and three months. A total of 50 nurses were screened, and 30 who met the inclusion criteria were enrolled and randomly assigned to the intervention (n = 15) or control (n = 15) group. Inclusion criteria included at least one year of experience in the same clinical setting and the provision of informed consent. Nurses with communication impairments that could interfere with participation were excluded.

The intervention consisted of six weekly online Balint-based group sessions lasting 45-50 minutes. Sessions followed the structure recommended by the International Balint Federation, including case presentation, exploration, group discussion, feedback, and closing phases. The first session included additional time to review study procedures and establish group rules and confidentiality. The control group continued routine work without receiving any additional psychosocial support.

The primary outcome was burnout, measured with the Maslach Burnout Inventory. The secondary outcome was communication skills, assessed with the Communication Skills Scale for Health Professionals. Both outcomes were measured at baseline, immediately after the intervention, and at one- and three-month follow-ups.

Data were collected electronically, and all participants provided informed consent online. Ethical approval was obtained from the relevant institutional ethics committee. This study contributes to the growing evidence supporting the use of Balint-based reflective group interventions to enhance nurses' psychosocial well-being and professional communication competencies.

DETAILED DESCRIPTION:
Nurses experience burnout as a response to prolonged exposure to stressors. Burnout significantly reduces nurses' capacity for therapeutic communication by weakening their empathy and active listening skills. Balint therapy is a reflective approach focused on the patient-nurse relationship. In Balint groups, nurses discover how to better manage challenging patient-nurse relationships and strive to improve their interpersonal relationships. Balint groups are particularly helpful in recognizing feelings and thoughts related to patients who are perceived as "difficult." Balint-based interventions are conducive to providing social support by creating a relatively safe atmosphere while respecting nurses' experiences. Furthermore, considering nurses' working conditions, Balint-based interventions are considered an easy-to-implement, time-efficient, and evidence-based approach.

The present study aims to measure the effect of Balint-based group intervention on burnout and communication skills among nurses. The research hypotheses are as follows: H0-1: There is no significant difference in burnout levels between the intervention and control groups. H0-2: There is no significant difference in communication skills between the intervention and control groups.

This study was conducted using a two-armed parallel group randomized controlled design with pre-test and post-test measurements, and follow-up assessments were performed at one and three months. Participants included nurses recruited using a purposive sampling method. The inclusion criteria were: (i) having worked as a nurse in the same clinical setting for at least one year and (ii) providing informed consent to participate. The exclusion criterion was the presence of a communication impairment that could hinder participation (e.g., hearing or speech disorder). The criteria for discontinuation from the study included: (i) voluntary withdrawal, (ii) missing at least two sessions, and (iii) incomplete or missing data on the study instruments. A total of 50 nurses were contacted by the research team and underwent eligibility screening. A total of 30 nurses who met the inclusion criteria were enrolled in the study, taking into account a potential dropout rate. The study was completed with a total of 30 nurses, 15 in the intervention group and 15 in the control group. Participants were randomly assigned to either the intervention or control group at a 1:1 ratio using simple randomization.

The primary outcome of the study is burnout, measured using the Maslach Burnout Inventory. Higher scores indicate higher levels of burnout. The secondary outcome is communication skills, measured using the Communication Skills Scale for Health Professionals, with higher scores indicating better communication skills. Both outcomes were assessed at baseline, after the intervention, and at one- and three-month follow-ups.

This study conducted from December 2024 to April 2025. Participating nurses received an online information form and a voluntary consent form. After reviewing the information, participants provided electronic consent. Only those who consented were included in the online intervention sessions.

Intervention group sessions were held once a week, each lasting 45-50 minutes, without disrupting nurses' rest periods or shift schedules. The intervention group was organized as a closed group. Session days were scheduled according to nurses' weekly work schedule. The groups were facilitated by two academically qualified researchers specializing in psychiatric nursing, each trained in psychotherapy techniques, including psychodrama and cognitive behavioral therapy. Sessions were conducted online in a quiet environment, with the screen layout designed to allow participants to see one another clearly. Nurses participated in Balint-based group counseling for six weeks. Post-tests were administered immediately after the final session (Session 6). The first follow-up assessment was conducted one month after the intervention, and the second follow-up assessment took place three months post-intervention.

The intervention in this study consisted of nurse-led group counseling based on the Balint approach. The primary objectives of a Balint group are to deepen understanding of the nurse-patient relationship, enhance nurses' awareness of their own emotions, thoughts, and behaviors within that relationship, and provide a supportive environment for participants. In this study, weekly sessions followed a structured format adapted from the recommendations of the International Balint Federation. The first session included an additional 30 minutes to explain the study's purpose and procedures, establish a confidentiality agreement, and clarify group rules and expectations (e.g., maintaining confidentiality, being respectful and non-judgmental, ensuring all members have an opportunity to speak, and attending sessions punctually). This preparation ensured that participants were fully prepared to engage in the intervention.

Phase 1 (Case Presentation): In each session, a different group member (the case presenter) shared a case involving a patient interaction that elicited intense or challenging emotions (e.g., distress, helplessness, frustration, anger). The case presenter elaborated on their feelings, thoughts, and behaviors regarding the situation, providing details about when, where, and how it occurred.

Phase 2 (Exploration): Group members asked questions to better understand the dynamics of the nurse-patient relationship in the case, while avoiding direct advice or criticism. The case presenter clarified ambiguous points and had the opportunity to explore their own experiences more deeply.

Phase 3 (Group Discussion): The group leader asked the case presenter to temporarily withdraw and remain silent during the discussion. Group members then discussed various aspects of the nurse-patient relationship, sharing their own feelings and perspectives. The group leader encouraged members to explore their emotions in depth and guided the discussion toward the dynamics of the nurse-patient relationship. By preventing criticism directed at the case presenter, the leader ensured a safe environment and effectively managed session time.

Phase 4 (Feedback): After the discussion, the case presenter rejoined the group to share new perspectives and emotional insights gained from the discussion. Group members then provided general evaluations of the process and highlighted their learning points.

Phase 5 (Closing): The group leader summarized the prominent themes that emerged during the session, offered a brief evaluation, and concluded the session in a structured manner.

Control group: Nurses in the control group continued their routine work schedules and did not receive any additional training or psychosocial support during the study period. Data collection instruments were administered to the control group concurrently with the intervention group. Because the nurses in the control group were employed at different hospitals and were unfamiliar with one another, the risk of information sharing between groups was minimized. After the study was completed, the control group was informed about the intervention; however, no additional counseling services were provided due to scheduling constraints related to their working hours.

Data were collected at baseline, immediately after the intervention, and at one- and three-month follow-ups. Sociodemographic characteristics of the groups were compared using chi-square tests or Fisher's exact tests for categorical variables and independent samples t-tests for continuous variables. A two-way mixed-design ANOVA was performed to examine between-group, within-time, and group × time interactions; the Bonferroni test was used for multiple comparisons. Paired sample t-tests were also used to compare pre-test and post-test scores in the intervention group. Effect sizes were reported using Cohen's d for within-group comparisons and partial eta-squared (η²) for the mixed ANOVA. Statistical significance was set at p < .05.

Ethical approval for this study was obtained from the Bilecik Seyh Edebali University Non-Interventional Clinical Research Ethics Committee (19.09.2024 - 280361). Prior to participation, nurses were provided with detailed information about the purpose of the study, the procedures to be performed, and the voluntary nature of participation. Informed consent was obtained electronically from all participants via an online consent form. Participants were assured of confidentiality, the right to withdraw from the study at any time, and that their personal information would not be shared.

ELIGIBILITY:
Inclusion Criteria:

* having worked as a nurse in the same clinical setting for at least one year
* providing informed consent to participate

Exclusion Criteria:

* presence of a communication impairment that could hinder participation (e.g., hearing or speech disorder)

Discontinuation Criteria:

* Voluntary withdrawal from the study
* Failure to attend at least two sessions
* Incomplete or missing data on the study instruments

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-12-20 (Actual); Primary Completion 2025-04-05 (Actual); Study Completion 2025-04-05 (Actual)

PRIMARY OUTCOMES:
Burnout (Maslach Burnout Inventory Total Score) | Baseline, immediately after the intervention (6 weeks), 1-month follow-up, and 3-month follow-up.
  Burnout will be assessed using the Maslach Burnout Inventory (MBI), a 22-item self-report scale measuring emotional exhaustion, depersonalization, and personal accomplishment. In this study, the personal accomplishment subscale will be reverse-coded so that higher total scores indicate higher levels of burnout. Scores range from 0 to 88. MBI is widely used to assess occupational burnout among healthcare professionals.

SECONDARY OUTCOMES:
Communication Skills (Communication Skills Scale for Health Professionals) | Baseline, immediately after the intervention (6 weeks), 1-month follow-up, and 3-month follow-up.
  Communication skills will be assessed using the Communication Skills Scale for Health Professionals (CSSHP), an 18-item self-report instrument evaluating communication attitudes and behaviors across four subscales. Items are scored on a 1-6 Likert scale, with higher scores indicating better communication skills. Total scores range from 18 to 108.

CONTACTS AND LOCATIONS:
Locations (1):
- Bilecik Şeyh Edebali University, Faculty of Health Sciences, Bilecik, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Huang L, Harsh J, Cui H, Wu J, Thai J, Zhang X, Cheng L, Wu W. A Randomized Controlled Trial of Balint Groups to Prevent Burnout Among Residents in China. Front Psychiatry. 2020 Feb 11;10:957. doi: 10.3389/fpsyt.2019.00957. eCollection 2019. PMID 32116808

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-09-19): https://cdn.clinicaltrials.gov/large-docs/19/NCT07278219/Prot_SAP_000.pdf
  • Informed Consent Form (2024-09-19): https://cdn.clinicaltrials.gov/large-docs/19/NCT07278219/ICF_001.pdf